CLINICAL TRIAL: NCT00613418
Title: Comparative Study of Safety and Efficacy of the SUPERA® Wire Interwoven Self-expanding Nitinol Stent and Currently Approved Stents for Patients With Iliac Lesions
Brief Title: Comparative Study Of Safety And Efficacy Of The SUPERA® Nitinol Stent - Iliac Artery
Acronym: I-WIN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study did not move forward due to change in clinical strategy
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Baim Institute for Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-1 - US
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: With de Novo or Restenotic Lesions in the Common and/or External Iliac Arteries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- single (Other): Historical control
  Interventions: Device: IDev SUPERA® Interwoven Self Expanding Nitinol Stent Peripheral Vascular System

INTERVENTIONS:
Device: IDev SUPERA® Interwoven Self Expanding Nitinol Stent Peripheral Vascular System — Interwoven, self-expanding nitinol stent system, including delivery system and stent

SUMMARY:
This is a prospective, multicenter, non-randomized, single-arm trial; the primary objective is to assess the comparability of the performance of the IDev SUPERA® nitinol stent to a rate derived from a meta-analysis of studies on iliac stents approved by FDA for treating subjects with de novo or restenotic lesions in the common and/or external iliac arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older and of legal age of consent.
2. Subject has lifestyle limiting claudication or rest pain (Rutherford-Becker scale 2, 3 or 4).
3. Subject has de novo or restenotic lesions in the common or external iliac artery.
4. Subject has single, bilateral or multiple target lesions that is (are) ≥ 50% stenosed by visual estimate.
5. The target lesion(s) can be successfully crossed with a guide wire and dilated.
6. The target segment of subject's lesion(s) is between 4 and 10 mm in diameter and less than 110 mm in length.
7. Subject has angiographic evidence of a patent femoral outflow artery in the target limb.
8. Subject has provided written informed consent.
9. Subject is able and willing to adhere to the required follow-up visits and testing through month 36.
10. Subject is able and willing to adhere to the required follow-up medication regimen

    -

Exclusion Criteria:

1. Presence of other non-target arterial lesions requiring treatment within 30 days of the procedure.
2. The target lesion(s) has adjacent, acute thrombus.
3. The target lesion(s) is highly calcified or was previously treated with a stent.
4. Subject has a pre-existing target iliac artery perforation or dissection of the target iliac artery prior to initiation of the IDev implant procedure.
5. Subject has an abdominal aortic aneurysm contiguous with the iliac artery target lesion. Subject has a pre-existing aneurysm or dissection of the target iliac segment.
6. Subject with aortic or iliac aneurysm that is likely to require repair within the next 9 months.
7. Subject has a post-surgical stenosis and anastomotic suture treatments of the target vessel.
8. Subject has a vascular graft previously implanted in the native iliac vessel.
9. Subject has tissue loss, defined as Rutherford-Becker classification category 5 or 6.
10. Subject is unable to accommodate ≥ 7 Fr cat
11. Subject has contrast agent hypersensitivity that cannot be adequately pre-medicated, has a hypersensitivity to nickel, or has intolerance to antiplatelet, anticoagulant, or thrombolytic medications.
12. Subject has history of neutropenia (WBC <3,000/mm3).
13. Subject has coagulopathy or thrombocytopenia (platelet count <80,000/ μL) that has not resolved or has required treatment in the past 6 months.
14. Subject has known bleeding or hypercoagulability disorder or significant anemia (Hb < 8.0 g/dL) that cannot be corrected.
15. Subject has the following laboratory values:

    1. international normalized ratio (INR) greater than 1.5,
    2. serum creatinine level greater than 2.5 mg/dL.
16. Subject requires general anesthesia for the procedure.
17. Subject is pregnant or plans to become pregnant during the study.
18. Subject has a co-morbid illness that may result in a life expectancy of less than 1 year.
19. Subject is participating in an investigational study of a new drug, biologic or device at the time of study screening. NOTE: Subjects who are participating in the long term follow-up phase of a previously investigational and now FDA-approved product are not excluded by this criterion.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of death | within 30 days post-procedure
Target site revascularization or restenosis | 9 months

SECONDARY OUTCOMES:
Major adverse events (MAEs) | 30 days
Device success (delivery and deployment of the study stent and retrieval of the delivery system) | During implantation procedure
Acute procedural success | immediately following stent deployment
Early and late clinical success (Rutherford-Becker improvement); ABI and TBI improvement; symptom based. | 30 days and 6, 9, and 12 months
Target vessel patency | 6, 9, 12, 24, and 36 months
Quality of Life questionnaire | baseline, 3 and 6 months